CLINICAL TRIAL: NCT00843011
Title: A Open-label, Randomized, Single-dose, 3-way Crossover Study to Investigate the Pharmacokinetics, Safety and Tolerability of 2 Different Formulations of Orvepitant and the Effect of Food in Healthy Volunteers.
Brief Title: Food and Relative Bioavailability Study
Acronym: Food/rel BA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 110355
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder
Keywords: formulation; safety and tolerability; pharmacokinetics; NK1 antagonist; effect of food
MeSH Terms: conditions — Depressive Disorder | interventions — orvepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Orvepitant 60 mg
  Interventions: Drug: Orvepitant

INTERVENTIONS:
Drug: Orvepitant — Orvepitant 60 mg, single dose. 2 different formulation. Formulation 2 is administered with and without food.

SUMMARY:
This study is an open-label, randomised, single dose study to determine the pharmacokinetics, safety and tolerability of 2 different formulations of orvepitant 60 mg and the effect of food in 15 Healthy Volunteers.

DETAILED DESCRIPTION:
Orvepitant is a highly potent and selective neurokinin-1 (NK1) receptor antagonist currently in development for the treatment of depression and anxiety.

This study is an open-label, randomised, single dose study to determine the pharmacokinetics, safety and tolerability of 2 different formulations of orvepitant 60 mg and the effect of food in 15 Healthy Volunteers. According to a cross over design, in three different occasions, each subject will receive the "old" formulation of orvepitant in fasted condition and the "new" formulation in fasted condition and after a FDA High-Fat Breakfast. Subjects will be screened within 21 days of first treatment. On each dosing occasion, subjects will be admitted to the clinic on Day-1 and will remain until Day 2; they will be also asked to return to the site 48 and 72 hours after each dosing for the PK blood sample collection. The wash-out period between each dosing occasion will be at least 5 days and subjects will be asked to return to the site 7-14 days after the administration of the last dose of orvepitant for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 18 and 65 years of age inclusive.
* A female subject is eligible to participate if she is of either non-childbearing potential or child-bearing potential and agrees to use one of the contraception methods
* No co-morbid Psychiatric Disorders as defined using the Mini International Neuropsychiatric Interview (M.I.N.I) scale.
* A 12-lead ECG at screening showed no abnormalities that in the opinion of the Principal Investigator will compromise safety in this study.

  -- Body weight ≥ 50 kg and BMI within the range 19.0 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent

Exclusion Criteria:

* As a result of any of the medical interview, physical examination or screening investigations the Physician Responsible considers the subject unfit for the study.
* The subject has a history of a drug or other allergy which in the opinion of the Physician Responsible contraindicates the participation in the study.
* Subjects with an unstable medical disorder or a disorder that would likely interfere with the action, absorption, distribution, metabolism or excretion of orvepitant, may pose a safety concern, or interfere with accurate assessment of safety.
* The subject has a current or recent (within six months) documented gastrointestinal disease; a history of malabsorption, oesophageal reflux, or irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn, or any surgical intervention (e.g. cholecystectomy) which would be expected to influence the absorption of drugs.
* History of psychiatric illness
* Any history of a clinically significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* Subject is consuming alcool or tobacco
* Subject is positive to Hepatitis B, C or HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08-28 (Actual); Primary Completion 2008-10-23 (Actual); Study Completion 2008-10-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic:parameters of orvepitant: tlag, tmax, Cmax, AUC(0-t), AUC (0-∞), t1/2. | 72 hours post dose.
Safety and tolerability endpoints will be evaluated by adverse event monitoring,laboratory values, cardiovascular monitoring | 5 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Verona, Veneto, Italy

REFERENCES:
- See also: Results for study 110355 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/110355?search=study&search_terms=110355#rs